CLINICAL TRIAL: NCT03391258
Title: Guided Bone Regeneration With L-PRF in the Atrophic Maxilla - A Pilot Clinical Trial
Brief Title: Guided Bone Regeneration With L-PRF in the Atrophic Maxilla - The GLAM Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implantology Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: II2015-06
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Bone Regeneration
Keywords: Maxilary atrophy; Leucocyte-platelet-rich-fibrin; bone resorption; autologous growth factors; guided-bone-regeneration; lip support
MeSH Terms: conditions — Bone Resorption | interventions — Bone Regeneration

STUDY DESIGN:
Intervention Model Description: To describe the dimensional changes (based on CBCT scans) occurred 12 months after implant placement and simultaneous regeneration with L-PRF and bovine bone graft in the aesthetic zone of atrophic maxillae in full arch implant supported rehabilitations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Regeneration with GLAM technique (Experimental): At the beginning of each surgery, a venipuncture will be performed, to obtain the L-PRF membranes. Also, two white topped tubes will be centrifuged for 3 minutes to obtain PRP. After implant placement, achieving a primary stability of at least 45 Ncm, the stiff bone-block (L-PRF membranes and PRP combined with bovine xenograft) will be used in the buccal plate of the pre-maxilla, to enhance bone volume in the esthetic area.
  Interventions: Procedure: Bone Regeneration with GLAM technique

INTERVENTIONS:
Procedure: Bone Regeneration with GLAM technique — Bone regeneration with GLAM technique in full arch implant supported rehabilitation

SUMMARY:
16 patients with severe resorbed maxillae referred to Implantology Institute® will be submitted to full arch surgery, with simultaneous implant placement and regeneration in the aesthetic zone, with the GLAM technique.

Informed consents and local ethical committee clearance will be obtained. Pre, post and 12 months' follow-up CBCT scans will be performed and 2 independent, calibrated operators will analyze the CBCT scans and mean bone values calculated. The distance from the nasopalatine canal to the center of each implant will be determined (4 different locations per patient, corresponding to implants 14; 11; 21; 24) and it will be the reference to other CBCTs. Implant length will be measured, from the neck (site 1) to the top and then a middle point will be assessed (site 2). Post-Surgical Volume (mm) will be determined from the most palatal point of cortical bone until the most buccal regenerated bone in each CBCT. Regenerated bone gain (mm) at post-op and at 1-year CBCTs will be calculated by the difference between pre and post-op or pre-op and 1 year CBCT measures, respectively. Regenerated Bone stability (%), defined as the percentage of regenerated bone at 12 months, will be calculated as the comparison between CBCT immediately after surgery and the CBCT at 12 months. Results will be presented as mean, with 95% CI.

DETAILED DESCRIPTION:
Patients with maxillary atrophy and loss of lip support are often a challenge in terms of prosthodontic rehabilitation and surgical approach due to the aesthetic changes and bone availability for implant placement.

In edentulous patients, with severe maxillary atrophy and an obvious loss of lip support, the anterior maxilla commonly exhibits a thin buccal bone plate which requires horizontal bone augmentation, since various authors have mentioned that a minimum 2mm of facial bone is required to prevent vertical bone resorption.

The scientific literature describes several techniques for these cases (such as collagen or titanium membranes, non-resorbable pins, use of xenografts, allografts or autogenous bone) but still, none is considered as the gold standard.

The simultaneous approach, where implant placement is coincident with graft procedures, is preferred by both patients and clinicians, since it reduces treatment time and cost. However, it can't be applied in every case, due to the need of proper implant stability.

A significant clinical interest has grown regarding the use of L-PRF for regeneration, solely or in combination with xenografts, given its ease of protocol preparation, economic advantages, less invasive technique (no need for donor sites) and biological properties. Also, L-PRF has been used around immediately placed implants to restore the anatomy loss and to speed up soft tissue wound healing. However, the use of enough L-PRF membranes seems to be crucial to obtain an optimal effect.

For this reason, the use of a Guided bone regeneration with L-PRF in the Atrophic Maxilla (GLAM) technique is suggested as a surgical approach in patients with maxillary atrophy and evident loss of lip support, where Guided bone regeneration is performed with the use of L-PRF membranes and xenograft to restore the buccal bone volume of the Atrophic Maxilla, simultaneously to implant placement.

Aim: The purpose of this clinical trial is to evaluate the dimensional changes in the aesthetic zone of resorbed maxillae (based on CBCT scans) occurred 12 months after implant placement and simultaneous regeneration with the GLAM technique.

SURGICAL PROTOCOL: At the beginning of each surgery, a venipuncture will be performed, and blood will be drawn into red topped tubes (BD Vacutainer ®, 10mL) and centrifuged at 2700 rpm (IntraSpin™ Centrifuge, Intra-Lock ®) for 12 minutes to obtain the L-PRF membranes. Also, two white topped tubes (BD Vacutainer ®, 9mL) will be centrifuged for 3 minutes to obtain PRP. Both L-PRF membranes and PRP will be prepared according to previously described protocols. After implant placement, achieving a primary stability of at least 45 Ncm, the stiff bone-block (L-PRF membranes and PRP combined with bovine xenograft) will be used in the buccal plate of the pre-maxilla, to enhance bone volume in the esthetic area. After handling and positioning the bone block, a minimum of 3 layers of L-PRF membranes will be placed over the graft, in order to enhance the soft tissue healing. In cases where primary closure is not achievable, the top layer of the membranes will be left exposed.

CBCT ANALYSIS: Pre-op, post-op and 12 months' follow-up CBCT scans will be performed. Two independent, calibrated operators will analyze the CBCT scans and mean values will be calculated.

The distance from the nasopalatine canal to the center of each anterior implant will be determined in the post-op CBCT, in the panoramic perspective, and this will be the reference value to the other CBCTs. Four different locations will be determined per patient, in the anterior region of the maxilla, delimited by the anterior border of the maxillary sinus. These locations corresponded to the former lateral incisors and first pre-molars positions.

In sagittal cuts of the CBCT, the implant length will be measured, from the neck (site 1) to the top. Afterwards, a middle point will be assessed (site 2). These sites are the reference for measurements of bone volume in all the CBCT scans. Both sites correspond to the most grafted areas of the implants when restoring the lip support, thus more susceptible to dimensional changes. The apical third of the implant is responsible for the palatal bone anchorage.

Considering the CBCT scans, the following variables will be measured in both sites 1 and 2:

Post-Surgical Volume (mm): determined from the most palatal point of cortical bone until the most buccal point of regenerated bone, perpendicular to the implant's long axis.

Regenerated Bone Gain (mm): measured at the post-op and the 12 months CBCT scans from the most palatal point of cortical bone until the most buccal point of regenerated bone, perpendicular to the implant's long axis. Calculated by the difference between pre and post-op CBCTs (regenerated bone gain at post-op) and by the difference between pre-op and 12 months CBCT measures (regenerated bone gain at 12 months).

Regenerated Bone Stability (%): defined as the percentage of regenerated bone at 12 months, compared to immediately after surgery.

The results will be presented as mean, with 95% CI. Paired or independent Student's t-Test or ANOVA were used in this analysis. Post hoc tests will be used as appropriate, and Alpha will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ≥18years of age, ASA I or ASA II patients

Exclusion Criteria:

* ASA III or ASA IV patients; uncontrolled diabetes, immunosuppressant medication, heavy smokers or pre-surgical infectious area next to the surgical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Changes in Regenerated Bone Gain (mm) | Pre-surgery, Baseline (0 days) and 12 month follow-up
  Measured at the post-op and the 12 months CBCT scans from the most palatal point of cortical bone until the most buccal point of regenerated bone, perpendicular to the implant's long axis. Calculated by the difference between pre and post-op CBCTs (regenerated bone gain at post-op) and by the difference between pre-op and 12 months CBCT measures (regenerated bone gain at 12 months).

SECONDARY OUTCOMES:
Regenerated Bone Stability (%) | Baseline (0 days) and 12 month follow-up
  defined as the percentage of regenerated bone at 12 months, compared to immediately after surgery
Post-Surgical Regenerated Bone Volume (mm) | Baseline (0 days)
  determined from the most palatal point of cortical bone until the most buccal point of regenerated bone, perpendicular to the implant's long axis

CONTACTS AND LOCATIONS:
Overall Officials: Duarte Marques, DDS, PhD, Principal Investigator — Implantology Institute; João Caramês, DDS, PhD, Study Director — Implantology Institute
Locations (1):
- Instituto de Implantologia, Lisbon, Portugal